CLINICAL TRIAL: NCT03786094
Title: An International, Phase 3, Multicenter, Randomized, Open- Label Trial Comparing Balixafortide in Combination With Eribulin Versus Eribulin Alone in Patients With HER2 Negative, Locally Recurrent or Metastatic Breast Cancer
Brief Title: Pivotal Study in HER2 Negative, Locally Recurrent or Metastatic Breast Cancer
Acronym: FORTRESS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was halted early due to failure to meet the primary endpoint.
Sponsor: Spexis AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POL6326-009
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Results first posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Breast Cancer; Locally Recurrent Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin; balixafortide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Eribulin (Active Comparator)
  Interventions: Drug: Eribulin
- Balixafortide + Eribulin (Experimental)
  Interventions: Drug: Eribulin; Drug: Balixafortide

INTERVENTIONS:
Drug: Eribulin — Eribulin alone
  Other Names: Eribulin Injection [Halaven]
Drug: Balixafortide — Balixafortide + Eribulin
  Other Names: POL6326
  Arms: Balixafortide + Eribulin

SUMMARY:
This is a phase 3, multicenter, open-label, randomized active-controlled, parallel group to investigate the efficacy, safety and tolerability of intravenous balixafortide given with eribulin versus eribulin alone in the treatment of HER2 negative, Locally Recurrent or Metastatic Breast Cancer.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed Breast cancer
* Metastatic Breast Cancer currently of stage IV disease or unresectable locoregionally recurrent breast cancer
* refractory to the most recent chemotherapy, documented by progression on or within six (6) months of therapy
* At least 14 days from the completion of any previous cancer therapy
* Adequate organ function
* Life expectancy of 3 months or more
* Willing and able to comply with the protocol and able to understand and willing to sign an informed consent

Key Exclusion Criteria:

* Previously treated with eribulin
* Peripheral neuropathy Grade ≥3
* Receipt of prior CXCR4 therapy
* Receipt of colony stimulating factors (CSFs) filgrastim, pegfilgrastim, or sargramostim, or radiation therapy within 14 days prior to study Day 1
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to balixafortide or eribulin or other agents used in the study
* Breast feeding or pregnant
* Patients with congestive heart failure, electrolyte abnormalities, bradyarrhythmias, known congenital long QT syndrome, QT interval corrected with Fridericia's formula (QTcF) ≥470 msec at baseline in the absence of bundle branch block, or currently taking drugs at known risk of prolonging the QT interval or causing torsades de pointes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2021-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: François Ringeisen, MD, Study Director — Polyphor Ltd.; Peter A Kaufman, MD, Principal Investigator — UVM medical center; USA; Javier Cortes, MD, Principal Investigator — IOB and VHIO; Spain
Locations (88):
- United States (28):
  - California Cancer Associates for Research and Excellence, Fresno, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCSF Mount Zion Cancer Center, San Francisco, California
  - Stanford Cancer Center South Bay, San Jose, California
  - Norwalk Hospital, Norwalk, Connecticut
  - Florida Cancer Specialists SOUTH - SCRI - PPDS, Fort Myers, Florida
  - Orlando Health, Orlando, Florida
  - Florida Cancer Specialists NORTH - SCRI - PPDS, St. Petersburg, Florida
  - Florida Cancer Specialists PAN - SCRI - PPDS, Tallahassee, Florida
  - Tallahassee Memorial HealthCare, Tallahassee, Florida
  - Florida Cancer Specialists EAST - SCRI - PPDS, West Palm Beach, Florida
  - University Cancer and Blood Center, LLC, Athens, Georgia
  - Piedmont Cancer Institute PC, Atlanta, Georgia
  - Orchard Healthcare Research Inc, Skokie, Illinois
  - Herbert-Herman Cancer Center, Sparrow Hospital, Lansing, Michigan
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Saint Luke's Cancer Institute 150 Entrance, Kansas City, Missouri
  - HCA Midwest Health - SCRI - PPDS, Kansas City, Missouri
  - Mercy Research Oncology, St Louis, Missouri
  - CHI Health St. Francis, Grand Island, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Queens Hospital Cancer Center, New York, New York
  - OHSU Knight Cancer Institute Hematology Oncology, Portland, Oregon
  - Magee Women's Hospital, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Tennessee City, Tennessee
  - University of Vermont Medical Center, Burlington, Vermont
  - West Virginia University Hospital, Morgantown, West Virginia
- Argentina (4):
  - Centro Polivalente de Asistencia e Investigación Clínica - CER San Juan, San Juan, Buenos Aires
  - Centro de Investigación Clínica - Clínica Viedma, Viedma, Río Negro Province
  - Sanatorio Parque de Rosario, Rosario, Santa Fe Province
  - CAIPO Centro para la atención integral del paciente oncológico, San Miguel de Tucumán
- Belgium (5):
  - Grand Hopital de Charleroi asbl, Charleroi, Hainaut
  - UZ Antwerpen, Antwerp
  - CHIREC Centre Hospitalier Interregional Edith Cavell, Brussels
  - UZ Gent, Ghent
  - CHU de Liège, Liège
- Brazil (7):
  - Centro de Oncologia Da Bahia, Bahia
  - Universidade de Caxias do Sul (IPCEM-UCS), Caxias do Sul
  - Liga Paranaense de Combate Ao Cancer - Hospital Erasto Gaertner, Curitiba
  - Hospital Sao Lucas Da Pontificia Universidade Catolica Do Rio Grande Do Sul (PUCRS), Porto Alegre
  - INCA Instituto Nacional De Cancer, Rio de Janeiro
  - Hospital de Base Da Faculdade de Medicina de São José Do Rio Preto, São José do Rio Preto
  - Clinica de Pesquisas e Centro de Estudos Oncologia Ginecologica e Mamaria Ltda, São Paulo
- Czechia (3):
  - Multiscan s.r.o - Onkologická ambulance, Hořovice
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice v Motole, Prague
- France (3):
  - Centre Léon Bérard Centre Régional de Lutte Contre Le Cancer Rhône Alpes, Lyon
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - EDOG - Institut Claudius Regaud - PPDS, Toulouse
- Italy (5):
  - Ospedale San Raffaele S.r.l. - PPDS, Milan, Lombardy
  - ASST di Monza - Azienda Ospedaliera San Gerardo, Monza, Milano
  - Azienda Ospedaliero Universitaria Di Bologna - Policlinico S Orsola Malpighi, Bologna
  - Azienda Ospedaliero Universitaria Policlinico Vittorio Emanuele, Catania
  - Azienda Ospedaliera Universitaria - Università degli studi della Campania "Luigi Vanvitelli", Napoli
- Russia (8):
  - LLC Evimed, Chelyabinsk
  - Krasnoyarsk Regional Oncology Center n.a. A.I. Kryzhanovskiy, Krasnoyarsk
  - Medical Center Tonus, Nizhny Novgorod
  - Budgetary Healthcare Institution of the Omsk region "Clinical Oncology Dispensary", Omsk
  - Evromedservis LCC, Pushkin
  - Mordovia State University, Saransk
  - Research Oncology Institute of Tomsk Scientific Center, Tomsk
  - Volgograd Regional Clinical Oncology Dispensary, Volgograd
- South Korea (4):
  - National Cancer Center, Goyang-si
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (12):
  - Hospital Universitario Virgen Macarena, Seville, Andalusia
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - ICO l'Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Quironsalud Barcelona, Barcelona, Catalonia
  - Hospital Universitari Arnau de Vilanova, Lleida, Catalonia
  - Hospital Universitario A Coruña, A Coruña
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital Universitario Vall D'Hebrón, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Ruber Internacional, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
- Taiwan (3):
  - Chi Mei Medical Center, Liouying, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
- Ukraine (4):
  - Municipal Institution City Clinical Hospital #4 of Dnipro City Council - PPDS, Dnipro
  - LLC Medical Center Family Medicine Clinic, Dnipro
  - Municipal Institution SubCarpathian Clinical Oncological Centre, Ivano-Frankivsk
  - CNCE of Lviv Regional Council Lviv Oncological Regional Therapeutical and Diagnostic Centre, Lviv
- United Kingdom (2):
  - Leicester Royal Infirmary, Leicester
  - Barts Cancer Institute, London

RESULTS

PARTICIPANT FLOW:
Groups:
- Balixafortide + Eribulin: Balixafortide: Balixafortide + Eribulin
  Balixafortide was administered as a single IV administration (5.5 mg/kg over at least 2 hours [±10 minutes]) on Days 1-3 and Days 8-10 of each 21-day cycle. Eribulin was administered IV at a dose of 1.4 mg/m2 over 2 to 5 minutes on Days 2 and 9 of each 21-day cycle.
- Eribulin Monotherapy: Eribulin was administered as a single IV administration (1.4 mg/m2 over 2-5 minutes) on Days 2 and 9 of each 21-day cycle.
Period: Overall Study
Arm/Group | Balixafortide + Eribulin | Eribulin Monotherapy
Started | 219 | 213
Overall Population (2nd Line+) | 219 | 213
3rd Line+ Population | 175 | 173
Completed | 10 | 11
Not Completed | 209 | 202

BASELINE CHARACTERISTICS:
Population: Overall Population (2nd Line+)
Groups:
- Eribulin Monotherapy: Eribulin: Eribulin alone
- Total: Total of all reporting groups
Arm/Group | Balixafortide + Eribulin | Eribulin Monotherapy | Total
Number analyzed (Participants) | 219 | 213 | 432
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (10.87) | 55.6 (11.07) | 55.0 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 218 | 211 | 429
  Male | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 9 | 19 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 197 | 174 | 371
  More than one race | 3 | 5 | 8
  Unknown or Not Reported | 5 | 8 | 13
Breast Cancer History [Mean (Standard Deviation); unit: years]
  Time since first diagnosis of breast cancer | 6.99 (6.096) | 7.21 (5.647) | 7.10 (5.873)
  Time since diagnosis of locally recurrent or metastatic disease | 2.96 (2.503) | 3.15 (2.427) | 3.05 (2.464)

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (2nd Line+ Population)
Description: To evaluate the efficacy of balixafortide + eribulin versus eribulin monotherapy on the primary endpoint of progression free survival (PFS). PFS, as assessed by the Independent Review Committee, defined as the time from the date of randomization to the earliest evidence of documented progressive disease or death from any cause. Patients who were alive without postbaseline assessments or without documented progressive disease, lost to follow-up, withdrew consent, started an anticancer therapy prior to observing a progressive disease or with an event documented after 2 or more missing tumor assessments were censored.
  PFS was evaluated according to RECIST v1.1 guidelines for complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD).
Time Frame: Patients received treatment until PD by RECIST v1.1 criteria was met or until one of the treatment discontinuation or study withdrawal criteria was met.
Population: Overall Population (2nd Line+)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Balixafortide + Eribulin | Eribulin Monotherapy
Number analyzed (Participants) | 219 | 213
months | 3.5 [2.8 to 4.2] | 4.0 [3.0 to 4.3]
Statistical Analysis 1: Comparison: Balixafortide + Eribulin vs Eribulin Monotherapy; Test type: Superiority; p = 0.4450, t-test, 2 sided; Hazard Ratio (HR) = 1.10, 96% CI 2-sided [0.85 to 1.41] — HR and associated 2-sided 96% CI are estimated by a Cox proportional hazards model stratified for randomization stratification factors including a fixed effect term for treatment arm

2. Primary Outcome: Progression Free Survival (3rd Line+ Population)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: 3rd Line+ Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Balixafortide + Eribulin | Eribulin Monotherapy
Number analyzed (Participants) | 175 | 173
months | 3.5 [2.8 to 4.2] | 4.0 [2.9 to 4.2]
Statistical Analysis 1: Comparison: Balixafortide + Eribulin vs Eribulin Monotherapy; Test type: Superiority; p = 0.6158, t-test, 2 sided; Hazard Ratio (HR) = 1.07, 96% CI 2-sided [0.81 to 1.41] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Overall Survival (3rd Line+ Population)
Description: To compare the overall survival (OS) between patients in the balixafortide + eribulin treatment arm versus eribulin monotherapy treatment arm. OS is defined as the time from date of randomization to date of death due to any cause. Patients who are lost to follow-up or are not known to have died at the time of data-cut-off for analysis or who do not have any follow up since randomization were censored.
Time Frame: The Investigator monitored the patient for OS status every 6 months (or more frequently) until: death, the patient withdrew consent to follow-up for survival, or until the patient was lost to follow-up (whichever occurred first).
Population: 3rd Line+ Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Balixafortide + Eribulin | Eribulin Monotherapy
Number analyzed (Participants) | 175 | 173
months | 11.0 [8.9 to 12.3] | 11.2 [8.9 to 14.0]
Statistical Analysis 1: Comparison: Balixafortide + Eribulin vs Eribulin Monotherapy; Test type: Superiority; p = 0.6126, t-test, 2 sided; Hazard Ratio (HR) = 1.08, 99.9% CI 2-sided [0.66 to 1.77]

ADVERSE EVENTS:
Time Frame: 5 months
Description: For the purposes of the clinical study report, a treatment-emergent adverse event (TEAE) was considered to have occurred at a similar rate between treatment arms if the percentage difference between arms was <5.0%. TEAEs were defined as AEs that occurred at or after administration of the first dose of any study treatment and through 30 days after the last dose of any study treatment.
Arm/Group | Balixafortide + Eribulin | Eribulin Monotherapy
All-Cause Mortality (participants affected / at risk) | 17/218 | 13/204
Serious Adverse Events (participants affected / at risk) | 62/218 | 54/204
Other Adverse Events (participants affected / at risk) | 214/218 | 197/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Balixafortide + Eribulin (N=218) | Eribulin Monotherapy (N=204)
Pneumonia (Infections and infestations) | 5 | 5
COVID-19 pneumonia (Infections and infestations) | 3 | 5
Sepsis (Infections and infestations) | 3 | 3
Device related infection (Infections and infestations) | 1 | 2
Erysipelas (Infections and infestations) | 1 | 1
Neutropenic infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Arthritis infective (Infections and infestations) | 0 | 1
Atypical pneumonia (Infections and infestations) | 1 | 0
Breast cellulitis (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0
Dermatitis infected (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 9
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Immune-mediated pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Disease progression (General disorders) | 5 | 5
General physical health deterioration (General disorders) | 1 | 1
Asthenia (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 5 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal compression (Gastrointestinal disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Brain oedema (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Metabolism and nutrition disorders) | 1 | 0
Metastases to central nervous system (Metabolism and nutrition disorders) | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Transaminases increased (Investigations) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Lens extraction (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Balixafortide + Eribulin (N=218) | Eribulin Monotherapy (N=204)
Alopecia (Skin and subcutaneous tissue disorders) | 59 | 62
Pruritus (Skin and subcutaneous tissue disorders) | 55 | 1
Rash (Skin and subcutaneous tissue disorders) | 23 | 0
Neutropenia (Blood and lymphatic system disorders) | 57 | 68
Anaemia (Blood and lymphatic system disorders) | 27 | 33
Leukopenia (Blood and lymphatic system disorders) | 18 | 20
Asthenia (General disorders) | 41 | 40
Fatigue (General disorders) | 29 | 35
Pyrexia (General disorders) | 11 | 13
Nausea (Gastrointestinal disorders) | 44 | 40
Diarrhoea (Gastrointestinal disorders) | 17 | 27
Stomatitis (Gastrointestinal disorders) | 25 | 11
Constipation (Gastrointestinal disorders) | 16 | 19
Vomiting (Gastrointestinal disorders) | 14 | 11
Neutrophil count decreased (Investigations) | 34 | 35
Alanine aminotransferase increased (Investigations) | 14 | 15
White blood cell count decreased (Investigations) | 12 | 16
Aspartate aminotransferase increased (Investigations) | 8 | 18
Neuropathy peripheral (Nervous system disorders) | 18 | 14
Dysgeusia (Nervous system disorders) | 12 | 10
Peripheral sensory neuropathy (Nervous system disorders) | 12 | 10
Infusion related reaction (Injury, poisoning and procedural complications) | 95 | 0
Decreased appetite (Metabolism and nutrition disorders) | 22 | 12

LIMITATIONS AND CAVEATS:
The trial was halted early due to failure to meet the primary endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT03786094/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-14): https://cdn.clinicaltrials.gov/large-docs/94/NCT03786094/SAP_001.pdf